CLINICAL TRIAL: NCT02843932
Title: Study of Subjective Perception of Motor Control During Psychogenic Disorders : Brain Mechanisms and Functional Imaging.
Brief Title: Subjective Perception of Motor Control During Psychogenic Disorders
Acronym: PERCMO-TNF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitment difficulties
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 38RC14.120*
Record Dates: First submitted 2015-05-12; First posted 2016-07-26 (Estimated); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Somatoform Disorders
Keywords: Somatoform; Psychogenic
MeSH Terms: conditions — Somatoform Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Psychogenic disorders (Experimental): Psychogenic movement disorders and seizures
  Interventions: Other: functional brain MRI

INTERVENTIONS:
Other: functional brain MRI — functional imagery during motor-perception tasks

SUMMARY:
The aim of this study is to reveal neurobiological bases of the motor control of conscious perception, thanks to new techniques of functional cerebral imaging (MRI), and potentials deteriorations connected to neuropsychiatric disorders like conversion disorder.

The Hospital University Center of Grenoble will provide patients from Neurology department, characterized with non psychogenic epileptic seizures and abnormal psychogenic movements, from conversive origin.

Subjects will be scanned by Magnetic Resonance Imaging during a motor paradigm inducing a perceptive conflict between two informations : proprioceptive information coming from the action (drawing) and visual information (draw's mark) that appears on the screen when there is movement.

DETAILED DESCRIPTION:
New results will be provided about brain mechanisms involved in motor control perception among healthy patients and patients suffering from functional neurologic symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Medical exam médical done before study participation
* Between 18 and 65 years
* Right-handed persons
* Conversion disorder based on DSM IV-R criterias
* Symptom affecting motor system, like abnormal movements (shivers, dystonia, parkinsonism, or problem when walking)

Exclusion Criteria:

* Subjects included in a clinical and/or therapeutic exeprimentation in progress
* People with MRI contraindications : prosthesis or metal implants, metallic teeth (dental) brace, pacemaker, IUD, possibility of pregnancy, claustrophobia
* Traitement médicamenteux psychotrope ou susceptible d'interférer avec le débit sanguin cérébral ou l'activité neuronale
* History of brain or disseminated and extendible lesions of white matter, of an other degenerative morbidity, a confusion or an insanity as well as serious deficits preventing language understanding.
* Alcohol ingestion
* Pregnant, parturient or breastfeeding women
* All other categories of protected persons

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-05-13 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Familiarization with the joystick. | 30 minutes
  HHSC-JOY-I from Current Designs. They are asked to trace a straight line.
Brain MRI | One hour and a half

CONTACTS AND LOCATIONS:
Overall Officials: Tiphaine Montagnon, Study Chair — DRCI, CHU GRENOBLE, FRANCE
Locations (1):
- Chu Grenoble, Grenoble, France

REFERENCES:
- [Background] Desmurget M, Grafton S. Forward modeling allows feedback control for fast reaching movements. Trends Cogn Sci. 2000 Nov 1;4(11):423-431. doi: 10.1016/s1364-6613(00)01537-0. PMID 11058820
- [Background] Wolpert DM, Ghahramani Z, Jordan MI. An internal model for sensorimotor integration. Science. 1995 Sep 29;269(5232):1880-2. doi: 10.1126/science.7569931.
- [Background] Sabes PN. The planning and control of reaching movements. Curr Opin Neurobiol. 2000 Dec;10(6):740-6. doi: 10.1016/s0959-4388(00)00149-5. PMID 11240283
- [Background] Rothwell JC, Traub MM, Day BL, Obeso JA, Thomas PK, Marsden CD. Manual motor performance in a deafferented man. Brain. 1982 Sep;105 (Pt 3):515-42. doi: 10.1093/brain/105.3.515. PMID 6286035
- [Background] Ghez C, Hening W, Gordon J. Organization of voluntary movement. Curr Opin Neurobiol. 1991 Dec;1(4):664-71. doi: 10.1016/s0959-4388(05)80046-7. PMID 1822314
- [Background] van Beers RJ, Baraduc P, Wolpert DM. Role of uncertainty in sensorimotor control. Philos Trans R Soc Lond B Biol Sci. 2002 Aug 29;357(1424):1137-45. doi: 10.1098/rstb.2002.1101. PMID 12217180
- [Background] Fourneret P, Jeannerod M. Limited conscious monitoring of motor performance in normal subjects. Neuropsychologia. 1998 Nov;36(11):1133-40. doi: 10.1016/s0028-3932(98)00006-2. PMID 9842759
- [Background] Carson AJ, Stone J, Warlow C, Sharpe M. Patients whom neurologists find difficult to help. J Neurol Neurosurg Psychiatry. 2004 Dec;75(12):1776-8. doi: 10.1136/jnnp.2003.032169. PMID 15548505
- [Background] Vuilleumier P, Chicherio C, Assal F, Schwartz S, Slosman D, Landis T. Functional neuroanatomical correlates of hysterical sensorimotor loss. Brain. 2001 Jun;124(Pt 6):1077-90. doi: 10.1093/brain/124.6.1077. PMID 11353724
- [Background] Cojan Y, Waber L, Carruzzo A, Vuilleumier P. Motor inhibition in hysterical conversion paralysis. Neuroimage. 2009 Sep;47(3):1026-37. doi: 10.1016/j.neuroimage.2009.05.023. Epub 2009 May 18. PMID 19450695
- [Background] Cojan Y, Vuilleumier P. Functional brain imaging of psychogenic paralysis during conversion and hypnosis
- [Background] Hallet M, cloninger CR, Fahn S, Halligan P, Jankovic J, Lang AE, Voon V Psychogenic movement disorders and other conversion disorders. Cambridge University Press 2011
- [Background] de Lange FP, Roelofs K, Toni I. Motor imagery: a window into the mechanisms and alterations of the motor system. Cortex. 2008 May;44(5):494-506. doi: 10.1016/j.cortex.2007.09.002. Epub 2007 Dec 23. PMID 18387583
- [Background] Blakemore SJ, Wolpert DM, Frith CD. Abnormalities in the awareness of action. Trends Cogn Sci. 2002 Jun 1;6(6):237-242. doi: 10.1016/s1364-6613(02)01907-1. PMID 12039604
- [Background] de Lange FP, Roelofs K, Toni I. Increased self-monitoring during imagined movements in conversion paralysis. Neuropsychologia. 2007 May 15;45(9):2051-8. doi: 10.1016/j.neuropsychologia.2007.02.002. Epub 2007 Feb 11. PMID 17367826
- [Background] Friston KJ, Holmes AP, Worsley KJ. How many subjects constitute a study? Neuroimage. 1999 Jul;10(1):1-5. doi: 10.1006/nimg.1999.0439. PMID 10385576
- [Background] Stone J, Carson A, Sharpe M. Functional symptoms in neurology: management. J Neurol Neurosurg Psychiatry. 2005 Mar;76 Suppl 1(Suppl 1):i13-21. doi: 10.1136/jnnp.2004.061663. No abstract available. PMID 15718216